CLINICAL TRIAL: NCT02482129
Title: A Multicenter, Randomized, Double-Masked, Active-Controlled Study to Evaluate the Safety and Efficacy of LME636 in Patients With Acute Anterior Uveitis
Brief Title: Proof of Concept Study to Evaluate Safety and Efficacy of LME636 in the Treatment of Acute Anterior Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LME636-2201
Record Dates: First submitted 2015-06-23; First posted 2015-06-26 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-07

CONDITIONS: Acute Anterior Uveitis
Keywords: Acute anterior uveitis; LME636
MeSH Terms: conditions — Uveitis, Anterior | interventions — Ophthalmic Solutions; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LME636 (Experimental): LME636 60 mg/mL ophthalmic solution, maximum drop frequency administered for 2 weeks, followed by a tapering for 1 week (Week 3) and 1 week of masked Vehicle administration (Week 4)
  Interventions: Drug: LME636 60 mg/mL ophthalmic solution; Drug: LME636 Vehicle
- Dexamethasone (Active Comparator): Dexamethasone 0.1% ophthalmic solution, maximum drop frequency administered for 2 weeks, followed by a tapering for 2 weeks (Weeks 3 and 4)
  Interventions: Drug: Dexamethasone 0.1% ophthalmic solution

INTERVENTIONS:
Drug: LME636 60 mg/mL ophthalmic solution
  Arms: LME636
Drug: Dexamethasone 0.1% ophthalmic solution
  Arms: Dexamethasone
Drug: LME636 Vehicle — Inactive ingredients used for masking purposes
  Arms: LME636

SUMMARY:
The purpose of the study is to determine whether topical ocular administration of LME636 60 mg/mL is efficacious in resolving the ocular inflammation in the anterior chamber (AC) associated with acute anterior uveitis (AAU).

DETAILED DESCRIPTION:
Eligible subjects will be randomized to LME636 or Dexamethasone in a 3:1 ratio at the time they present to the trial site with the AAU flare and will enter treatment for 28 full days. Subjects with worsening disease from Visit 2/Day 4 onward or subjects without improvement after 14 days of treatment will be discontinued from treatment, unmasked and treated with a rescue regimen at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Diagnosis of non-infectious AAU in at least 1 eye.
* Anterior chamber cell score of 2+ or 3+ as per Standardization of Uveitis Nomenclature (SUN) in at least one eye.
* Able to communicate well with the Investigator, to understand and comply with the requirements of the study.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of child-bearing potential unwilling to use effective contraception methods as defined in the protocol.
* AC cell score of 4+ (SUN) or hypopyon.
* Onset of anterior uveitis more than 2 weeks prior to enrollment in the study.
* Presence of intermediate-, posterior-, or panuveitis in either eye.
* Administration of stable doses >10 mg daily systemic prednisone or corticosteroids as described in the protocol.
* Recurrent corneal abrasion or ulceration in either eye (past or present).
* Tuberculosis (past or present).
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Scientist NIBR, Alcon, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 10 study centers located in the United States.
Pre-assignment Details: Of the 45 enrolled, 2 subjects were exited as screen failures prior to randomization and 4 subjects were randomized, but not treated. This reporting group includes all randomized subjects, as treated. Note: One subject randomized to LME636 was treated with dexamethasone instead.
Period: Overall Study
Arm/Group | LME636 | Dexamethasone
Started | 32 | 11
Treated, as Randomized | 30 | 9
Completed | 26 | 9
Not Completed | 6 | 2
Not completed — Adverse Event-prior to treatment | 0 | 1
Not completed — Withdrawal by subject-prior to treatment | 0 | 1
Not completed — Unable to draw blood-prior to treatment | 1 | 0
Not completed — Criteria not met-prior to treatment | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Criteria not met | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and treated subjects, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | LME636 | Dexamethasone | Total
Number analyzed (Participants) | 29 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (17.20) | 55.6 (16.02) | 54.5 (16.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders at Day 15
Description: Response was defined as a two-step decrease or more from baseline in Anterior Chamber (AC) Cell Grade as per Standardization of Uveitis Nomenclature (SUN). Baseline was defined as the measurement taken before drug administration on Day 1. Subjects receiving rescue treatment on or before Day 15 were considered non-responders. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Day 15
Population: This analysis population includes all subjects who received any study drug, had at least 1 post-baseline efficacy assessment, had no critical protocol deviations, and had a valid determination of response status for the primary endpoint (Per Protocol Analysis Set).
Measure: Count of Participants; unit: Participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 25 | 10
Participants | 14 | 9

2. Primary Outcome: Mean Best Corrected Visual Acuity (BCVA) at Each Visit
Description: Visual Acuity (VA) with the subject's best spectacles or other visual corrective devices was measured using an Early Treatment of Diabetic Retinopathy Study (ETDRS) or Snellen visual acuity chart and reported in letters read correctly. An increase (gain) in letters read indicates improvement. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Day 4, Day 8, Day 15, Day 22, Day 29
Population: This analysis population includes all subjects who received any study drug (Safety Analysis Set). Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
letters
  Baseline | 71.1 (14.58) | 77.2 (14.69)
  Day 4: number analyzed (Participants) | 28 | 10
  Day 4 | 70.5 (13.92) | 77.9 (12.94)
  Day 8: number analyzed (Participants) | 27 | 10
  Day 8 | 72.1 (13.62) | 76.8 (11.50)
  Day 15: number analyzed (Participants) | 26 | 10
  Day 15 | 74.1 (10.11) | 77.1 (11.82)
  Day 22: number analyzed (Participants) | 25 | 10
  Day 22 | 74.5 (10.41) | 78.2 (11.31)
  Day 29: number analyzed (Participants) | 25 | 10
  Day 29 | 73.8 (11.70) | 79.2 (11.23)

3. Primary Outcome: Mean Intraocular Pressure (IOP) at Each Visit
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry or Tonopen and reported in millimeters mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Day 4, Day 8, Day 15, Day 22, Day 29
Population: Safety Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
mmHg
  Baseline (Day 1) | 15.2 (5.09) | 15.5 (4.12)
  Day 4: number analyzed (Participants) | 28 | 10
  Day 4 | 14.8 (3.74) | 15.3 (3.47)
  Day 8: number analyzed (Participants) | 27 | 10
  Day 8 | 14.1 (3.40) | 16.1 (3.51)
  Day 15: number analyzed (Participants) | 26 | 10
  Day 15 | 14.0 (3.38) | 16.0 (5.06)
  Day 22: number analyzed (Participants) | 25 | 10
  Day 22 | 14.6 (3.14) | 17.0 (4.57)
  Day 29: number analyzed (Participants) | 25 | 10
  Day 29 | 15.5 (4.72) | 16.3 (4.40)

4. Primary Outcome: Number of Subjects With Increase From Baseline in Slit Lamp Parameters at Any Post-Treatment Visit
Description: Slit-lamp biomicroscopy (examination) was performed to evaluate the anterior segment of the eye, including lids/lashes, conjunctiva, cornea, anterior chamber (cells and flare), iris, and lens. Ocular signs were categorized as Aqueous Flare, Aqueous Inflammatory Cell Grade, Keratic Precipitates, Lens, Limbal Injection, Status of Lens, Peripheral Anterior Synechia, and Posterior Synechia. An increase indicates worsening. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Day 4, Day 8, Day 15, Day 22, Day 29
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
participants
  Aqueous Flare | 9 | 1
  Aqueous Inflammatory Cell Grade | 4 | 1
  Keratic Precipitates | 4 | 0
  Lens | 0 | 0
  Limbal Injection | 7 | 0
  Status of Lens | 0 | 0
  Peripheral Anterior Synechia | 1 | 1
  Posterior Synechiae | 8 | 1

5. Primary Outcome: Number of Subjects With an Increase From Baseline in Dilated Fundus Parameters at Any Post-Treatment Visit
Description: The dilated fundus examination was performed to evaluate the health of the vitreous, optic disc, retinal vessels, macula, and retinal periphery. An increase indicates worsening. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Day 4, Day 8, Day 15, Day 22, Day 29
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
participants
  Macula | 2 | 0
  Optic Nerve | 1 | 0
  Retina | 1 | 0
  Vitreous | 4 | 0

6. Secondary Outcome: Number of Subjects With IOP Change From Baseline to Last On-Treatment Assessment
Description: IOP was assessed using Goldmann applanation tonometry or Tonopen and reported in mmHg. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Up to Day 29
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
Participants
  Increase > 30 mmHg | 0 | 0
  Increase 11-30 mmHg | 1 | 0
  Increase 6-10 mmHg | 0 | 2
  -5 mmHg Decrease - 5 mmHg Increase | 25 | 8
  Decrease 6-10 mmHg | 1 | 0
  Decrease 11-30 mmHg | 2 | 0
  Decrease > 30 mmHg | 0 | 0

7. Secondary Outcome: Mean Change From Baseline in BCVA at Each Visit
Description: Visual Acuity (VA) was measured with the participant's best spectacles or other visual corrective device in place using an ETDRS or Snellen visual acuity chart. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Day 4, Day 8, Day 15, Day 22, Day 29
Population: Safety Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
letters
  Baseline (BL) | 71.1 (14.58) | 77.2 (14.69)
  Change from BL at Day 4: number analyzed (Participants) | 28 | 10
  Change from BL at Day 4 | -0.1 (9.74) | 0.7 (5.40)
  Change from BL at Day 8: number analyzed (Participants) | 27 | 10
  Change from BL at Day 8 | 0.0 (12.84) | -0.4 (6.19)
  Change from BL at Day 15: number analyzed (Participants) | 26 | 10
  Change from BL at Day 15 | 2.1 (9.53) | -0.1 (3.73)
  Change from BL at Day 22: number analyzed (Participants) | 25 | 10
  Change from BL at Day 22 | 2.8 (9.10) | 1.0 (5.06)
  Change from BL at Day 29: number analyzed (Participants) | 25 | 10
  Change from BL at Day 29 | 2.1 (10.36) | 2.0 (5.37)

8. Secondary Outcome: Time-to-Response
Description: Time-to-Response was defined as the number of days from baseline to the first scheduled visit when a two-step decrease or more from baseline in AC Cell Grade (as per SUN) was observed. Time-to-Response is reported as number of subjects presenting time-to-response by visit. Only one eye contributed to the analysis.
Time Frame: Baseline (Day 1), Up to Day 15
Population: Per Protocol Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 25 | 10
Participants
  Day 4 | 9 | 7
  Day 8 | 5 | 2
  Day 15 | 1 | 0
  Non-Responder | 10 | 1

9. Secondary Outcome: Use of Rescue Treatment
Description: Use of rescue treatment is presented as the number of subjects with first use of rescue treatment by visit. Subjects receiving rescue medication were not considered withdrawn and the collection of data continued after discontinuation of study treatment. Only one eye contributed to the analysis.
Time Frame: Day 4, Day 8, Day 15
Population: Per Protocol Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 25 | 10
Participants
  Day 4 | 3 | 0
  Day 8 | 3 | 0
  Day 15 | 0 | 0
  No Rescue | 19 | 10

10. Secondary Outcome: Mean Serum Concentration of Total LME636 at Each Visit
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method. Concentrations below the limit of quantification (BLQ), defined as 0.25 ng/mL, were reported as NA with no imputation for missing data.
Time Frame: Baseline (Day 1), Day 4, Day 8, Day 15, Day 22, Day 29
Population: This analysis population includes all subjects who received investigative product (IP) and had at least 1 evaluable serum sample following IP exposure.(Pharmacokinetics Analysis Set). Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LME636
Number analyzed (Participants) | 29
ng/mL
  Day 1 | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.
  Day 4: number analyzed (Participants) | 25
  Day 4 | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.
  Day 8: number analyzed (Participants) | 22
  Day 8 | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.
  Day 15: number analyzed (Participants) | 20
  Day 15 | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.
  Day 22: number analyzed (Participants) | 20
  Day 22 | 0.2510 (0.31237)
  Day 29: number analyzed (Participants) | 19
  Day 29 | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation.

11. Secondary Outcome: Number of Subjects With Anti-LME636 Antibodies Present at Each Visit
Description: Serum samples were collected and assessed for anti-LME636 antibodies. Samples collected from subjects in the LME636 dose group were analyzed for anti-LME636 antibodies. For subjects in the dexamethasone group, only the samples collected on Day 1 (ie, prior to the start of treatment) were analyzed for anti-LME636 antibodies.
Time Frame: Day 1, Day 4, Day 8, Day 15, Day 22, Day 29
Population: This analysis population includes all subjects with available immunogenicity data and no protocol deviations with relevant impact on the data (Immunogenicity Set).
Measure: Count of Participants; unit: Participants
Arm/Group | LME636 | Dexamethasone
Number analyzed (Participants) | 29 | 10
Participants
  Day 1 | 5 | 3
  Day 4: number analyzed (Participants) | 26 | 0
  Day 4 | 5 |
  Day 8: number analyzed (Participants) | 23 | 0
  Day 8 | 6 |
  Day 15: number analyzed (Participants) | 20 | 0
  Day 15 | 11 |
  Day 22: number analyzed (Participants) | 20 | 0
  Day 22 | 17 |
  Day 29: number analyzed (Participants) | 20 | 0
  Day 29 | 18 |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 35 days). AEs are reported as pretreatment, treatment-emergent, and posttreatment.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from participants and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- LME636: All subjects exposed to LME636 ophthalmic solution
- Dexamethasone: All subjects exposed to Dexamethasone ophthalmic solution
- Posttreatment: All subjects from the conclusion of treatment until exit from the study
Arm/Group | Pretreatment | LME636 | Dexamethasone | Posttreatment
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/29 | 0/10 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/29 | 0/10 | 0/39
Other Adverse Events (participants affected / at risk) | 0/45 | 13/29 | 6/10 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=45) | LME636 (N=29) | Dexamethasone (N=10) | Posttreatment (N=39)
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=45) | LME636 (N=29) | Dexamethasone (N=10) | Posttreatment (N=39)
Anterior chamber cell (Eye disorders) | 0 | 4 | 1 | 0
Anterior chamber flare (Eye disorders) | 0 | 3 | 0 | 0
Ciliary muscle spasm (Eye disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 2 | 0 | 0
Eye pain (Eye disorders) | 0 | 4 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 3 | 1 | 0
Iris adhesions (Eye disorders) | 0 | 3 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 3 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.